CLINICAL TRIAL: NCT05007119
Title: "Cupping Therapy Combined With Conventional PT Improves Pain and Health Related Quality of Life Among Female Patients of Low Back Pain''
Brief Title: "Cupping Therapy Combined With Conventional Physical Therapy Improves Pain and Health Related Quality of Life Among Female Patients of Low Back Pain''
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/9
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2020-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Cupping Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): It includes participants receiving conventional physical therapy for low back pain female patients for a period of 6 months.
  McKenzie extension exercise Protocol Moist Heat Pack for 10 mins McKenzie Extension Protocol Sequence
  Static:
  1. Lying Prone
  2. Lying prone in extension
  3. Sustained extension
  4. Posture correction
     Dynamic:
  5. Extension in lying
  6. Extension in lying with clinician overpressure
  7. Extension mobilization
  8. Extension in standing
  Interventions: Procedure: Mckenzie Extension Protocol
- Experimental Group (Experimental): Group (A) Involves participants receiving cupping therapy along with conventional physicla therapy for a period of 6 months .
  Moist Heat Pack for 10 mins McKenzie Extension Exercise Protocol
  Interventions: Procedure: Mckenzie Extension Protocol; Procedure: Cupping

INTERVENTIONS:
Procedure: Mckenzie Extension Protocol — Moist Heat Pack for 10 mins McKenzie Extension Protocol Sequence
  Static:
  1. Lying Prone
  2. Lying prone in extension
  3. Sustained extension
  4. Posture correction
     Dynamic:
  5. Extension in lying
  6. Extension in lying with clinician overpressure
  7. Extension mobilization
  8. Extension in standing
Procedure: Cupping — Cupping with blood letting
  Arms: Experimental Group

SUMMARY:
A randomized control trial will be done on diagnosed Low Back Pain patients in Fauji Foundation Hospital Rawalpindi. There is a growing interest and demand in the field of Complementary And Alternative Medicine(CAM), nowadays .The purpose of the study is to determine the effects of cupping therapy combined with conventional physical therapy to exercise to lower the pain and improve the health related quality of life of the patient using the modified SF - 36 scale. The conventional physical therapy includes hot pack placed on the low back region for ten minutes, interferential current therapy was used which has four round electrodes measuring 2.75 inches placed on the desired area(low back) waveform used was IFC- 4p , having a carrier frequency of 4000 Hz and a frequency of 80/150 Hz, vector scan was off , the intensity was increased manually according to the capacity of the patient and the treatment time was 15 minutes, strenghtening exercises such as william flexion were done once in the rehabilition center and patient was given a home plan to follow twice daily with 15 repitions each.

DETAILED DESCRIPTION:
Experimental Group (A) = This group will receive cupping therapy every month combined with conventional physical therapy whhich includes hot pack , interferential therapy and streghtening exercises for back and their outcomes wi;; be measured at baseline and at the end of 6th month treatment..

Control group (B) =this group will not receive cuppping therapy , only conventional Physical therapy will be given and their outcomes will be observed at the baseline and then after treatment of 06 months.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study within the community using the VAS scale.

A printed questionnaire will be provided to the parents after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

This study will make people become aware of their current physical fitness level, so the lifestyle behaviors can be modified if needed, in order to improve their quality of life This study will help create awareness among the people, it is not only economically accessible but also have very little chances of side effects This study will open new doors for researchers to do long term studies on different types of pain with different exercise types.

ELIGIBILITY:
Inclusion Criteria:

1. Female population of age between 30 to 50 years.
2. Female patients with diagnosed low back pain.

Exclusion criteria:

Female population with cardiological, neurological, circulatory and orthopedic problems opens wounds or bone fractures.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain | 8 weeks
Health Related Quality of life | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No